CLINICAL TRIAL: NCT06796595
Title: Perioperative Medical Program to Optimize Nerve Regeneration After Robot-assisted Laparoscopic Neurolyses of Pudendal and/or Inferior Cluneal Nerves for Chronic Neuralgias: Results After 1-year Follow-up
Acronym: REGEN
Status: Recruiting | Type: Observational
Sponsor: UBOSGA (Other)
Responsible Party: Sponsor
Other Study IDs: UBOSGA 2025/01
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Pudendal Neuralgia; Neuralgia
MeSH Terms: conditions — Pudendal Neuralgia; Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pudendal and inferior cluneal neuralgias are responsible for chronic pelvicperineal pain. These two neuralgias are associated in approximately 25% of cases. In the event of failure of first-line multimodal medical treatment, a mini-invasive robot-assisted laparoscopic decompression can be proposed. These surgeries carry the risk of neurapraxia, leading to a temporary increase in neuropathic pain and numbness in the nerve sensitive area, a motoric or neurovegetative disturbance (pudendal).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Patients presenting a pudendal and/or inferior cluneal neuralgias with failure of the medical treatment
* Patient having given consent after reading the information note

Exclusion Criteria:

* Inoperable patients (contraindications to anesthesia or surgery) surgical contraindications)
* Person deprived of liberty or under guardianship
* Person under court protection
* Pregnant or breast-feeding woman
* Minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This cohort study is a pilot study to evaluate the 1-year effectiveness of a perioperative medical program on the characteristics of neuropathic pain related to postoperative neurapraxia, following robot-assisted laparoscopic neurolyses of the pudendal and inferior cluneal nerves
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-01-23 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the 1-year effectiveness of a perioperative medical program on the characteristics of neuropathic pain related to postoperative neurapraxia, following robot-assisted laparoscopic neurolyses of the pudendal and inferior cluneal nerves | Pré-operatively, and then post-operatively : every day the first month, then once a week until the 4th month then at 1 year year after surgery
  Numeric pain scale (0 "no pain" to 10 "maximal pain")

SECONDARY OUTCOMES:
Report all complications during the follow-up | 2 days, 4 months, 1 year after surgery
  Complications are evaluated with Clavien-Dindo classification (Grade I to V(death))
Evaluate the effect of the surgical technique on anxiety | Pré-operatively, 2 days, 4 months, 1 year after surgery
  Anxiety is evaluated with STAI (State Trait Anxiety Inventory-form) (anxious personality since STAI score 51 for women, and score 61 for men)
Evaluate the effect of the surgical technique on depression | Pré-operatively, 2 days, 4 months, 1 year after surgery
  Depression is evaluated with Beck inventory (mild to moderate depression since score 10, moderate depression since score 19, severe depression since score 30)
Evaluate the effect of the surgical technique on post-traumatic stress syndrome | Pré-operatively, 2 days, 4 months, 1 year after surgery
  Post-traumatic stress syndrome is evaluated with PCL-5 (post-traumatic stress disorder checklist with a PTSD since score 38
Evaluate the impact on quality of life | Pré-operatively, 2 days, 4 months, 1 year after surgery
  Quality of life is evaluated with SF-36 (36-item Short Form Health Survey)

CONTACTS AND LOCATIONS:
Locations (1):
- UBOSGA, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No